CLINICAL TRIAL: NCT03216330
Title: Endometriosis Deep Dyspareunia and Central Sensitization
Brief Title: Dyspareunia and Central Sensitization
Status: Completed | Type: Observational
Sponsor: BC Women's Hospital & Health Centre (Other)
Responsible Party: Principal Investigator, Paul Yong, Principal Investigator and Research Director, BC Women's Centre for Pelvic Pain and Endometriosis., BC Women's Hospital & Health Centre
Other Study IDs: H16-02903
Record Dates: First submitted 2017-07-09; First posted 2017-07-13 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis; Central Sensitisation; Dyspareunia
Keywords: Quantitative sensory test (QST); Deep dyspareunia; Electronic Thimble Algometer
MeSH Terms: conditions — Endometriosis; Dyspareunia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: * Consented to participate in the Data Registry (H16-00264) prior to their physician appointment at the BC Women's Health Centre.
  * New or re-referred to the BC Women's Health Centre for Pelvic Pain and Endometriosis.
  * Endometriosis (previously surgically diagnosed, or current endometrioma, or current nodule)
  * Willing and committed to indicating pain scores and menstrual data on a REDCap survey every day for 6 weeks after the test date.
  * At least 18 years old
  Interventions: Other: No Intervention
- Control: * Reproductive aged female with no suspected or diagnosed endometriosis.
  * Have not experienced any sexual pain scores over 4/10 on a 11-point numeric rating scale, as determined on an online questionnaire prior to test day.
  * At least 18 years old
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no treatment intervention. We are assigning measurement tools such as the Electronic Thimble Algometer for QST and questionnaires to both groups.

SUMMARY:
Background: Endometriosis affects 10% of reproductive aged females, and can have a negative impact on sexual quality of life. Endometriosis can cause pelvic pain with deep penetration during intercourse, as well as other sexual and non-sexual pains. This study will allow us to determine if an increase in sexual pain is related to central sensitization.

Purpose: The purpose of this study is to determine if there is an association between the severity of sexual pain and central sensitization in women with endometriosis.

Measurement tools: Data will be collected from the Clinic's Data Registry, an online questionnaire, a quantitative sensory test (QST) to measure pain-pressure threshold (PPT) as a marker of central sensitization, and daily entry to an online survey.

Primary Hypothesis: Central sensitization (measured by lower pain-pressure threshold) will be associated with an increased severity of deep dyspareunia, as well as a tenderness of the bladder/pelvic floor and depression, in women with endometriosis.

DETAILED DESCRIPTION:
Background:

Endometriosis results from the presence of endometrial cells growing abnormally outside the uterus and affects approximately 10% of reproductive-aged females. Endometriosis can be associated with various types of pain such as: dysmenorrhea (painful cramps with menses), deep dyspareunia (pelvic pain with deep penetration during intercourse), dyschezia (painful bowel movements) and chronic pelvic pain. Few studies have explored the association between endometriosis and deep dyspareunia resulting in a limited understanding of how to treat deep dyspareunia. Deep dyspareunia is defined as pelvic pain with deep penetration and occurs in 50% of women with endometriosis at some time in their sexual lives. Deep dyspareunia has been shown to lower or cease intercourse, thus lowering self-esteem and resulting in negative effects on sexual functioning and interpersonal relationships.

A potential contributor to deep dyspareunia in women with endometriosis that is largely under-researched is the concept of central sensitization. Central sensitization is an amplification of nociceptive signaling that may result from prolonged pain causing sensitization of the dorsal horn neurons, which results in hyperalgesia (increased response to pain) and allodynia (response to pain when there normally would not be). A recent study, comparing cross-sectional data from suspected or surgically diagnosed endometriosis patients, suggested that bladder and pelvic floor tenderness may be markers of central sensitization. However, the linkage between the indirect markers of central sensitization and the presence of central sensitization requires confirmation. This link can be assessed through validated quantitative sensory testing (QST). Likewise, the association between central sensitization and deep dyspareunia may also be confirmed through QST. QST is an objective measurement tool to determine the presence and/or degree of sensory disturbances, by detecting the alterations in nociceptive pathways. For example, a low pain-pressure threshold (i.e., increased pain sensation) at healthy unaffected areas, as measured by QST, indicates central sensitization.

Purpose: To determine if deep dyspareunia is associated with central sensitization in women with endometriosis.

Research Question: Is deep dyspareunia associated with central sensitization assessed by decreased pain-pressure threshold?

Objectives:

Primary Objective:

1. Examine the association between central sensitization and severity of deep dyspareunia.

Secondary Objectives:

1. Examine the association between central sensitization and severity of non-sexual pains and Endometriosis Health Profile (EHP-30) scores.
2. Examine the association between central sensitization and tenderness of the bladder and pelvic floor (determined by physician on physical exam).
3. Examine the association between central sensitization and psychological measures (assessed by validated questionnaires).

   Research Hypotheses:

   Primary Hypothesis: Central sensitization (measured by pain-pressure threshold) is associated with an increased severity of deep dyspareunia, as well as a tenderness of the bladder/pelvic floor and depression, in women with endometriosis.

   Secondary Hypothesis: Women with endometriosis will have greater central sensitization (indicated by a lower pain-pressure threshold) than women without endometriosis.

   Setting: The Pelvic Pain and Endometriosis program at the BC Women's Health Centre uses an interdisciplinary approach to managing pain, including: physiotherapy for bladder and pelvic floor, surgical intervention, pain education and medical management. This program addresses multiple factors influencing pain through multiple approaches, as opposed to the traditional approach of surgical removal of the endometriosis to resolve the pain alone.

   Design: This study is a longitudinal, prospective cohort study, involving cases and controls.

   Primary Outcome: Severity of deep dyspareunia (0-10 numeric rating scale)

   Secondary Outcomes: Severity of superficial dyspareunia, severity of non-sexual pains, and psychological questionnaire scores

   Main Independent Variables: Central sensitization measured by pain-pressure threshold (PPT) determined through QST

   Study Population: The case population includes women who have consented to the Data Registry (H16-00264) and who are newly or re-referred to the BC Women's Centre for Pelvic Pain and Endometriosis, and who have regardless of the severity of deep dyspareunia, either: 1) previous surgical diagnosis of endometriosis or 2) current ovarian endometrioma cyst or 3) current endometriosis nodule.

   Sample Size: 30 cases and 15 controls.

   Recruitment and Data Collection prior to Test date:

   Cases:

   • At the end of their appointment with one of the endometriosis specialists at the BC Women's Centre for Pelvic Pain and Endometriosis, the physician will ask the patient if they are interested in learning more about this research study (if the physician deems them acceptable to be included based on screening of inclusion and exclusion criteria), and if so, will tell them a research assistant may call them.

   • A poster introducing the study will also be available in the clinic waiting rooms.

   • During a phone conversation, research team will remind the potential case participant that they have consented to the data registry, and consent to this study allows us access to analyze their data registry data. Verbal consent will be given if the potential case participant would like to participate, and a test appointment will be booked.

   • Case participants will sign the consent form in-person at the beginning of the test day appointment.

   Control:

   • Recruitment of the control group will be done by poster advertisement, as well as an in-person information session at the BC Women's Hospital. If they are interested in the study, potential participants will be asked to contact the research team to learn more about the study.

   • Research team will provide the potential control participant with a copy of the consent form (in person or by email). Each potential control participant will be advised to carefully read the consent form, and to contact the research team with any questions about the information contained in the consent form.

   • If the control participant expresses interest in the study after reading the consent form, a link to access the screening questions will be sent to them.

   • Criteria will be assessed by screening questions. If the participants are eligible based on the screening questions then they will be asked if they would like to consent to the study (online consent). This online consent allows access to the data from the screening questions. If they are not eligible, or do not consent to the study their screening questions will not be analyzed. If the control participant consents online they will be asked to complete additional questions (height, etc.).

   • Research team will receive an email once the control participant has consented online, and will contact the participant to book an appointment.

   • On the test day, the consent participants will sign the same consent form in-person to consent to the testing procedures.

   Procedures for Data Collection (on Test day)

   Questionnaire:

   Case and Control:

   • An online questionnaire will collect data such as: score of sexual and non-sexual pains, first day of last menstrual period,etc. The pelvic pain questions asked on this online questionnaire are modified from the Brief Pain Inventory Short Form. This questionnaire will be filled out online during the test appointment.

   Quantitative Sensory Testing (QST):

   Case and Control:
   * After the questionnaire has been completed, the participants will undergo QST to measure their pressure-pain threshold (PPT), the point where the sensation of pressure has changed to the sensation of pain. Before testing begins, it will be made clear that the participants can withdraw from the study even during the procedure if they find it too uncomfortable.
   * The PPT data will be written down on a paper copy with the unique study ID, and entered into an encrypted excel file.
   * The observation made by this QST is that a lower PPT is suggestive of increased central sensitization.

   Feedback Questionnaire:

   Case and Controls:

   • After the participant's PPT has been measured, they will be given an anonymous feedback form to assess the procedure mechanisms and specifications, as well as comfort level before, during and after testing. This will allow investigators to adjust any necessary procedure details to create a more comfortable environment/test for future participants.

   Procedures for Data Collection (after Test day)

   Online Survey:

   Cases only:
   * Case participants will be asked to record study data daily for six weeks after their scheduled test date.
   * The data collected, will allow for daily prospective pain scores, rather than retrospective recollections of pain scores.

   Participants without email addresses will have the opportunity to complete the surveys on a printed out copy (given to them on the appointment day) and mail/bring in-person to the Centre at the end of the 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Case:

  * Consented to participate in the Data Registry (H16-00264) prior to their physician appointment at the BC Women's Health Centre.
  * New or re-referred to the BC Women's Health Centre for Pelvic Pain and Endometriosis.
  * Endometriosis (previously surgically diagnosed, or current endometrioma, or current nodule)
  * Willing and committed to indicating pain scores and menstrual data on a REDCap survey every day for 6 weeks after the test date.
  * At least 18 years old
* Control:

  * Reproductive aged female with no suspected or diagnosed endometriosis.
  * Have not experienced any sexual pain scores over 4/10 on a 11-point numeric rating scale, as determined on an online questionnaire prior to test day.
  * At least 18 years old

Exclusion Criteria:

- Case and Control:

* Fibromyalgia.
* Severe and enduring psychological illness(es) affecting cognition (e.g., bipolar disorder, schizophrenia etc.).
* Currently pregnant or breastfeeding.
* Have a peripheral or central neurological disorder.
* Have diabetes mellitus or neuropathic pain.
* Do not speak English.
* Have had previous physical trauma (ex. Surgery) to the test site(s) (deltoid muscle in the shoulder, and first dorsal interosseous muscle).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Tertiary care centre (BC Women's Health Centre for Pelvic Pain and Endometriosis) for case participants.
  Community sample for control participants.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Deep dyspareunia score | Case and Control:1 day (same day as the QST testing date), and Case only: daily for 6 weeks after QST testing date
  Self reported on an 11-point numeric rating scale (10 being worst pain imaginable)

SECONDARY OUTCOMES:
Superficial Dyspareunia score | Case and Control:1 day (same day as the QST testing date), and Case only: daily for 6 weeks after QST testing date
  Self reported on an 11-point numeric rating scale (10 being worst pain imaginable)
Dysmenorrhea score | Case and Control:1 day (same day as the QST testing date)
  Self reported on an 11-point numeric rating scale (10 being worst pain imaginable)
Bladder and pelvic floor tenderness | Case only: 1 day (one week before the QST testing date)
  Yes/No determined through physical exam by a gynecologist
Chronic pelvic pain score | Case and Control:1 day (same day as the QST testing date), and Case only: daily for 6 weeks after QST testing date
  Self reported on an 11-point numeric rating scale (10 being worst pain imaginable)
Depression | Case only: 1 day (one week before the QST testing date)
  Patient Health Questionnaire (PHQ-9)
Anxiety | Case only: 1 day (one week before the QST testing date)
  Generalized Anxiety Disorder (GAD-7)
Catastrophizing | Case only: 1 day (one week before the QST testing date)
  Pain Catastrophizing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yong, MD/PhD, Principal Investigator — BC Children's and Women's Hospital
Locations (1):
- BC Children's and Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No